CLINICAL TRIAL: NCT01001611
Title: An Evaluation of Glycemic Control Effects of Mono Therapy CKD-501 in Patients With Type 2 Diabetes Mellitus: A 24-week, Multi Center, Randomized, Double-blind, Parallel-group, Placebo Control, Therapeutic Confirmatory Study
Brief Title: An Evaluation of Glycemic Control Effects of Mono Therapy CKD-501 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CKD-19DM09B; 19DM09B
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; glitazone; Type II Diabetes; Hypolipidemic; oral hypoglycemic agent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lobeglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CKD-501 0.5mg (Experimental)
  Interventions: Drug: CKD-501 0.5mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CKD-501 0.5mg — 0.5 mg/tablet, orally, 1 tablet once daily for 24 weeks or 52 weeks (If extension study)
  Other Names: Lobeglitazone
  Arms: CKD-501 0.5mg
Drug: Placebo — Indistinguishable tablet from CKD-501, Orally, 1 tablet once daily for 24 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate and confirm hypoglycemic efficacy and safety of CKD-501 as mono therapy in patients with type 2 diabetes treated once daily for 24 weeks in comparison to placebo.

DETAILED DESCRIPTION:
Diabetes Mellitus is classified into type 1 diabetes and type 2 diabetes mellitus according to the causes of diabetes onset and the treatment of symptoms.

In type 2 diabetes, the combination of insulin resistance and insulin deficiency is working. Diabetes mellitus causing many complications and hospitalization is one of chronic metabolic disorder and diabetes mortality rate has been gradually increasing percentage.

CKD-501 is highly selective peroxisome proliferator-activated receptor-gamma agonist that decreases insulin resistance in the periphery and liver resulting in increased insulin-dependent glucose disposal and decreased hepatic glucose output. In vivo, It demonstrates that CKD-501 improves even more glycemic and lipid control in comparison to rosiglitazone and pioglitazone.

The aim of this phase 3 study was to evaluate the efficacy and safety of CKD-501 once daily for 24 weeks as a monotherapy in type 2 diabetes mellitus. Furthermore, the extension study for additional 28 weeks is designed to confirm long term safety of CKD-501 as an oral hypoglycemic agent.

ELIGIBILITY:
Inclusion Criteria:

* Type Ⅱ diabetes mellitus
* Between 18 years and 80 years old
* The patient who has been taking oral hypoglycemic agent since 3 months with HbA1c 6.5 to 9% at screening test or who is drug naive or stopped taking oral hypoglycemic agent more then 3 months with HbA1c 7 to 10% at screening test
* BMI between 21kg/㎡ and 40kg/㎡
* Diagnosis of type Ⅱ diabetes before 3 months
* C-peptide level is over 1.0 ng/ml
* Condition for female having contraception methods, surgical sterilization or menopause
* Condition for male agreeing to use of recommendatory and appropriate contraception method
* Agreement with written informed consent

Exclusion Criteria:

* Type I diabetes, gestational diabetes or secondary diabetes
* Treatment with insulin or thiazolidinediones within 60 days
* Fasting Plasma Glucose level is over 250 mg/dl
* Triglyceride level is 500 mg/dl and over
* Uncontrollable hypertension(Although treat with antihypertension agent, systolic blood pressure greater than 140 mmHg and diastolic blood pressure greater than 90 mmHg)
* History of myocardial infarction, heart failure, cerebral infarction, hematencephalon or unstable angina within 6 months
* Severe hepatic dysfunction: AST, ALT, Total bilirubin, ALP level over or equal to 2.5 times as high as upper normal limit(UNL)
* Severe renal dysfunction: Renal failure or serum creatinine greater than 30% normal limit
* Anemia for any reason
* Needs treatment for acute disease, uncontrolled other diseae or diabetic complications
* Abnormality of thyroid function(out of normal TSH range )
* History of proliferative diabetic retinopathy
* In treatment concomitant drug having severe risk drug interaction with investigational drug
* History of cancer within 5 years
* History of drug abuse or alcoholism
* Hepatitis B Antigen(HBsAg) test is positive
* Treatment systemic or inhalant corticosteroids within 1 month prior to Screening
* Patient who have experience such as hypersensitivity reaction, serious adverse event or no effect by treatment with glitazones
* Fertile women who not practice contraception with appropriate methods
* Pregnant women or nursing mothers
* Has a contraindication to treatment investigational drug from the medical and psychogenic side
* An impossible one who participates in clinical trial by legal or investigator's decision
* Participated in other trial within 4 weeks
* Participating in other trial at present

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin (HbA1c) | 24 weeks

SECONDARY OUTCOMES:
Change from baseline in HbA1c target achievement rate (HbA1c<7%) | 24 weeks
Change from baseline in lipid parameters (Total cholesterol, Triglycerides(TG), LDL-C, HDL-C, Small Dense LDL-C, Free fatty acid(FFA), Apo-AⅠ/B/C Ⅲ) | 24 weeks
Evaluate safety of CKD-501 from physical exam, vital sign, laboratory test, adverse event and so on | 24 weeks or 52 weeks
Change from baseline in glycemic parameters (Fasting Plasma Glucose, C-peptide, Homeostasis Model Assessment of Insulin Resistance(HOMA-IR), Homeostasis Model Assessment of β-cell function(HOMA-β), Quantitative Insulin Check Index(QUICKI)) | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dongseop Choi, Study Chair — The Korea University Anam Hospital
Locations (9):
- South Korea (9):
  - The Inje University Busan-Paik Hospital, Busan
  - Soon Chun Hyang University Cheonan Hospital, Cheonan
  - The Hanyang University Medical Center, Gyeonggi-do
  - Wonju Severance Christian Hospital, Kangwon-Do
  - The Hallym University Medical Center, Seoul
  - The Inje University Sanggye-Paik Hospital, Seoul
  - The Korea University Anam Hospital, Seoul
  - The Kyung Hee University Medical Center, Seoul
  - The Seoul National University Bundang Hospital, Seoul

REFERENCES:
- [Derived] Kim SG, Kim DM, Woo JT, Jang HC, Chung CH, Ko KS, Park JH, Park YS, Kim SJ, Choi DS. Efficacy and safety of lobeglitazone monotherapy in patients with type 2 diabetes mellitus over 24-weeks: a multicenter, randomized, double-blind, parallel-group, placebo controlled trial. PLoS One. 2014 Apr 15;9(4):e92843. doi: 10.1371/journal.pone.0092843. eCollection 2014. PMID 24736628